CLINICAL TRIAL: NCT01731197
Title: Comparison of the Satiating Effects of Differentially Processed Isolated Soy Proteins
Brief Title: Satiating Effects of Isolated Soy Proteins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DuPont Nutrition and Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GIL-1245
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Weight Management
Keywords: obesity, isolated soy protein, satiety, food intake
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Test ISP-10 (Experimental): 10 grams of the test ISP will be consumed as a dry-blended beverage
  Interventions: Dietary Supplement: Dry-Blended Beverage
- Test ISP-20 (Experimental): 20 grams of the test ISP will be consumed as a dry-blended beverage
  Interventions: Dietary Supplement: Dry-Blended Beverage
- Control ISP-10 (Active Comparator): 10 grams of the control ISP will be consumed as a dry-blended beverage
  Interventions: Dietary Supplement: Dry-Blended Beverage
- Control ISP-20 (Active Comparator): 20 grams of the control ISP will be consumed as a dry-blended beverage
  Interventions: Dietary Supplement: Dry-Blended Beverage

INTERVENTIONS:
Dietary Supplement: Dry-Blended Beverage

SUMMARY:
Proteins are known to be more satiating than the other macronutrients; however, the type and amount of protein needed to induce a significant effect on satiety (fullness between meals) is sometimes difficult to determine. In this study, 2 differentially processed isolated soy proteins will be tested for satiety using subjective visual analogue scales. The amount of food consumed following intake of the isolated soy proteins will be measured 3 hours after consuming the proteins. The hypothesis is that differentially processed isolated soy proteins will show unique satiety responses.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 20 and 30 kg/m2
* Age between 18-65y
* Unrestrained eater (score<12)
* Regularly consume 3 meals per day
* Moderate exercise (eg running, aerobics classes, other sports activities) of no more than 7 hours per week

Exclusion Criteria:

* use of drugs that influence carbohydrate or lipid metabolism (eg. hypoglycemic agents, antibiotics taken less than 6 weeks before study entry, glucocorticoids, anti-diarrheal medication, weight loss medication, and anti-diabetic medication)
* presence of any significant disease (eg gastrointestinal diseases, diabetes, a CVD event less than 12 weeks from study entry, current hepatic disease, etc)
* use of special dietary treatments within 4 weeks of study (eg weight loss diet, extremely high or low carbohydrate/protein/fat diet, use of meal replacements more than once a day)
* use of supplements within 1 week of study (does not include vitamin supplements or supplements which are routinely taken and were initiated 4 weeks before the study and which will be continued during the study period)
* restrained eater (score>12)
* weight change (absolute body weight change of ≥ 10%) within the previous 6 weeks
* alcohol intake >2 drinks/day
* food allergies of any kind
* swallowing difficulties
* exercising more than 7 hours per week

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Subjective Satiety | 3 hours
  Measure subjective satiety using visual analogue scales

SECONDARY OUTCOMES:
Ad Libitum Food Intake | 30 minutes
  At the end of 3 hours after consuming test diets, measure the amount of food consumed for 30 mins

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wolever, MD, Principal Investigator — Glycemic Index Laboratories, Inc; Alexandra Jenkins, PhD, Principal Investigator — Glycemic Index Laboratories, Inc
Locations (1):
- Glycemic Index Laboratories, Toronto, Ontario, Canada